CLINICAL TRIAL: NCT01860391
Title: Salivary Levels of Fluoride and Silver 7 Days After Treatment With Diammine Silver Fluoride
Brief Title: Silver and Fluoride Salivary Levels After the Application of Silver Fluoride
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Peruana Cayetano Heredia (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single
Other Study IDs: 0000060585
Record Dates: First submitted 2013-05-20; First posted 2013-05-22 (Estimated); Last update posted 2013-05-22 (Estimated); Status verified 2013-05

CONDITIONS: Dentin Hypersensitivity
Keywords: Silver; Fluoride; Diammine Silver Fluoride; Saliva
MeSH Terms: conditions — Dentin Sensitivity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Application of Diammine SIlver Fluoride (Experimental): GROUP A (6 TEETH): 18 mcL will be expressed from a Hamilton syringe into a dappen dish, and then a single preweighed microbrush will be used to apply the material to the tooth surface after drying with cotton gauze. The 6 teeth will be treated consecutively until all the material in the dappen dish will be used. Then the brush will be reweighed to establish the non-applied amount.
  GROUP B (28 TEETH) Measure out 3 mcL X number of teeth present into dappen dish. Procedure is the same.
  Interventions: Device: Diammine Silver Fluoride

INTERVENTIONS:
Device: Diammine Silver Fluoride — Diammine SIlver Fluoride will be applied to teeth. The levels of silver and fluoride in saliva will be measure up to 7 days
  Other Names: Silver FLuoride; Saforide

SUMMARY:
The aim of the study is to measure salivary fluoride and silver levels up to 7 days post-treatment.

The participants will be 6 healthy adults. They will be given a fluoride free toothpaste to use the day before the study and all during the study.

3 participants will have 6 teeth treated (Group A).3 participants will have 28 teeth treated each on the facial aspect (Group B).

On day 0, the participant will be given 25 ml of de-ionized fluoride free water to swish in the mouth and spit the entire contents into a 50 ml collection tube. This will be done 3 times.

On day 0, 10 minutes after the rinsing and spitting, the participant will provide a unstimulated salivary sample into a universal collection tube until 5 ml are collected. The tubes with saliva will be stored on ice and then frozen at -20oC for transfer to the lab at the University of Washington.

On Day 0, Isolation and application of silver fluoride.

The quadrant will be isolated with cotton rolls, and surrounding gingiva will be covered with petroleum jelly to provide additional protection.

After application, participant will be given 25 ml of fluoride free water to rinse as in 1 above and water collected. This will be done 10 times.

DAY 1-6 Salivary Collection

Measures: Fluoride will be measured using standard fluoride electrode analysis (Martinez-Mier et al., 2011). Silver will be measured using Inductively Coupled Plasma-Mass Spectrometry (EPA 6020a Rev.1 2007) at the University of Washington

DETAILED DESCRIPTION:
Aim: to measure salivary fluoride and silver levels up to 7 days post-treatment. Based on extrapolation of the study by Vasquez and colleagues (2012), it is hypothesized that 7-day levels in the clinical study will not exceed baseline values.

Participants: 6 healthy adults of either sex, 21+ years old, who do not have gingivitis but who have generalized gingival recession >1mm, 3 subjects must have at least 28 teeth.

Participants will be given a fluoride free toothpaste to use the day before the study and all during the study. Participants will be reminded not to use fluoride toothpaste or other fluoride products and to avoid fish and tea.

No toothbrushing or eating at all within an hour of any visit

Design: Observational study with each participant as his/her own control.

3 participants will 6 treated (Group A).3 participants will have 28 teeth treated each on the facial aspect (Group B). Teeth with anterior fillings or decay at the gingival where staining would show will not be treated.

Day 0 Procedures:

1. On day 0, the participant will be given 25 ml of de-ionized fluoride free water to swish in the mouth and spit the entire contents into a 50 ml collection tube. This will be done 3 times.
2. On day 0, 10 minutes after the rinsing and spitting, the participant will provide a unstimulated salivary sample. The individual will be instructed to swallow once, and allow saliva to pool in the mouth without swallowing, and then periodically spit the saliva into a universal collection tube until 5 ml are collected. The tubes with saliva will be stored on ice and then frozen at -20oC for transfer to the lab at the University of Washington.
3. Day 0, Isolation and application of silver fluoride.

   GROUP A (6 TEETH): 18 mcL will be expressed from a Hamilton syringe into a dappen dish, and then a single preweighed microbrush will be used to apply the material to the tooth surface after drying with cotton gauze. The 6 teeth will be treated consecutively until all the material in the dappen dish will be used. Then the brush will be reweighed to establish the non-applied amount.

   GROUP B (28 TEETH) Measure out 3 mcL X number of teeth present into dappen dish. Procedure is the same.

   Application of silver fluoride. The quadrant will be isolated with cotton rolls, and surrounding gingiva will be covered with petroleum jelly to provide additional protection.
4. Day 0, after application, participant will be given 25 ml of fluoride free water to rinse as in 1 above and water collected. This will be done 10 times.

   DAY 1-6 Salivary Collection
5. Days 1-6, collection a single salivary sample at same time each day.

Procedure: Ten minutes before collection (on days 1-6), each individual will be given 100 ml of de-ionized fluoride free water to rinse the mouth and swallow to increase hydration. The individual will be instructed to swallow once, and allow saliva to pool in the mouth without swallowing, and then periodically spit the saliva into a universal collection tube until 5 ml are collected. The tubes with saliva will be stored on ice and then frozen at -20oC for transfer to the lab at the University of Washington.

Measures: Fluoride will be measured using standard fluoride electrode analysis (Martinez-Mier et al., 2011). Silver will be measured using Inductively Coupled Plasma-Mass Spectrometry (EPA 6020a Rev.1 2007).

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least one canine or premolar
* Patients with Dentin hypersensitivity
* Patients with healthy gingiva

Exclusion Criteria:

* Patients taking any of these medication: antidepressivem anticonvulsive, antihistaminic, antihypertension, antihemetic, antiespasmodic.
* Pregnancy
* Patients under radiation therapy
* Patients under chemotherapy
* Patients with alterations of salivary glands like Sjogren syndrome or Diabetes Mellitus with Xerostomia
* Patients with sensitivity to silver or other ions of heavy metals

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 6 (Actual)
Dates: Start 2012-12; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Silver and Fluoride levels in saliva | 7 days
  The daily fluoride and silver levels in saliva will be determined after the application of silver fluoride.

CONTACTS AND LOCATIONS:
Overall Officials: Adriana Romo, DDS, Principal Investigator — Universidad Peruana Cayetano Heredia